CLINICAL TRIAL: NCT00435175
Title: Acute Effects of Estradiol on Lipolysis in Subcutaneous Adipose Tissue and Muscle Assessed by Microdialysis and Tissue Biopsies
Brief Title: Acute Metabolic Effects of Estradiol
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: 2002-0242
Record Dates: First submitted 2007-02-13; First posted 2007-02-14 (Estimated); Last update posted 2007-02-14 (Estimated); Status verified 2007-02

CONDITIONS: Postmenopause
Keywords: Estradiol; Lipolysis; Estrogen receptor; Adrenergic receptors; UCP2; Postmenopausal women
MeSH Terms: interventions — Estradiol

INTERVENTIONS:
Drug: estradiol

SUMMARY:
Estradiol promotes and maintains the typical female phenotype characterized by subcutaneous fat accumulation. There is evidence to suggest that this effect relies on the ability of estradiol to increase the amount of anti-lipolytic α2A-adrenergic receptors, but whether this requires long-term exposure to estradiol or is the result of an immediate effect is not clear. Objective: To study acute effects of a single dose (4 mg) of 17β-estradiol on regional and systemic lipolysis.

DETAILED DESCRIPTION:
Estradiol affects muscle and fat distribution, and thereby lipid metabolism. A reduction in muscle power is seen after menopause, readily counteracted by female hormone therapy (HT). Treatment with HT through months to previously untreated postmenopausal women, or hormone replacement therapy (HRT) to women with Turner syndrome, increases muscle mass and reduces fat mass. HT in postmenopausal women furthermore prevents fat accumulation and increases lipoprotein lipase activity and lipolysis to an extent comparable to premenopausal women. In contrast, it has also been shown that estradiol may actually attenuate lipolysis during basal as well as catecholamine stimulated conditions. In addition, one study found whole body fat metabolism to be lower during treatment with estradiol than without, and reduced lipolysis is present in postmenopausal women during treatment with estradiol, along with an increased number of α-adrenergic receptors and a decreased number of β-adrenergic receptors.

It is not clear whether the lipolytic effect of estradiol happens acutely or is dependent on chronic exposure. Moreover, regional differences in the pharmacodynamics of estradiol have not been assessed. Finally, effects on skeletal muscle have never been examined.

The purpose of the present study was 1) by microdialysis to quantify the regional production of glycerol in two tissues (muscle and fat), and in two regions (abdominal and femoral). 2) To quantify the whole-body lipolytic effect of estradiol, and 3) in biopsies to study intracellular mechanisms behind the action of estradiol.

ELIGIBILITY:
Inclusion Criteria:

* Postmenopausal women assessed by FSH and estradiol levels
* Not taking any drugs
* Non-smokers

Exclusion Criteria:

* Obesity (BMI>30)

Ages: 45 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 8
Dates: Start 2005-06; Study Completion 2006-07

PRIMARY OUTCOMES:
Regional lipolysis assessed by microdialysis
Systemic lipolysis assessed by the isotope dilution technique
Lipoprotein lipase activity
Adrenergic receptor mRNA expression

SECONDARY OUTCOMES:
Estrogen receptor mRNA expression
UCP2 mRNA expression

CONTACTS AND LOCATIONS:
Overall Officials: Lars C Gormsen, MD, Principal Investigator — Aarhus University, Clinical Institute
Locations (1):
- Medical Research Laboratories, Aarhus, Denmark